CLINICAL TRIAL: NCT02454894
Title: Optimization Lumbar Puncture In Children
Acronym: OLPIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the reason that not all participants agree to have anesthesia and postoperative management at the same time
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Gang Liu, Chief physician/Professor, Beijing Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20150206
Record Dates: First submitted 2015-03-13; First posted 2015-05-27 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-05

CONDITIONS: Spinal Puncture Complications
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): no anesthesia; postoperative management
  Interventions: Procedure: postoperative management
- Group 2 (No Intervention): no anesthesia; lying without the pillow and fasting water and food for four hours after lumbar puncture
- Group 3 (Experimental): surface anesthesia with lidocaine; postoperative management
  Interventions: Drug: lidocaine; Procedure: postoperative management
- Group 4 (Experimental): surface anesthesia with lidocaine; lying without the pillow and fasting water and food for four hours after lumbar puncture
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine — surface anesthesia with lidocaine
  Arms: Group 3; Group 4
Procedure: postoperative management — lying without the pillow for half an hour after lumbar puncture
  Arms: Group 1; Group 3

SUMMARY:
The study is carried out in a prospective randomized controlled way. In the context of informed understanding from parents, compared with traditional process(no anesthesia; lying without the pillow and fasting water and food for four hours after lumbar puncture), randomly select lidocaine surface anesthesia and postoperative management (lying without the pillow for half an hour after lumbar puncture) . All children will be evaluated by the FLACC(The face,legs,activity,cry,consolability behavioral tool) scale to assess the degree of pain during and after lumbar puncture. Lumber puncture time, success rate and any postoperative condition will be recorded and analyzed.A questionaire about the operation for all parents and children will be investigated in order to establish an optimized lumbar puncture management process.

DETAILED DESCRIPTION:
The purpose of this study is to establish an optimized lumbar puncture management process on the basis of fully understanding of parents and children. An improved process consisting of painless lumbar puncture (LP),less postoperative complications and comfortable LP will be anticipated.

ELIGIBILITY:
Inclusion Criteria:

* children with indications of lumbar puncture;
* voluntarily signed the informed consent

Exclusion Criteria:

* topical anesthetic skin allergies;
* skin infection in lumbar puncture site;
* severe intracranial hypertension;
* unstable vital signs;
* coagulopathy;
* intracranial hemorrhage and occupying;
* low back pain;
* headache and low back pain before lumbar puncture;
* past headache after lumbar puncture;
* mental retardation, neuropsychiatric symptoms;
* children could not immediately act after the lumbar puncture(such as disturbance of consciousness or suffering from underlying diseases or drainage);
* the case with repeated puncture in one operation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Postoperation complications include headache, backache, vomit, cerebral hernia, allergy | up to five days postoperation

SECONDARY OUTCOMES:
Composite measure of Vital signs include heart rate, pulse, blood pressure and respiration. | up to four hours postoperation
degree of adaptability | intraoperative
  evaluated by the FLACC(The face,legs,activity,cry,consolability behavioral tool) scale
time of lumbar puncture | intraoperative
number of puncture | intraoperative
success rate | intraoperative
comfort degree | up to four hours postoperation
  evaluated by the FLACC(The face,legs,activity,cry,consolability behavioral tool) scale
whether bad memories exist or not | up to four hours postoperation
  A questionaire about the operation for all parents and children will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Liu, MD, Principal Investigator — Beijing Childrens' Hospital